CLINICAL TRIAL: NCT06915363
Title: Pivotal, Prospective, Randomized, Controlled, Multicenter Clinical Trial of BioPoly® Partial Resurfacing Knee Implant for Treatment of Focal Cartilage Lesions of the Distal Femur
Brief Title: BioPoly® Partial Resurfacing Knee Implant IDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BioPoly LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1150117
Record Dates: First submitted 2025-03-24; First posted 2025-04-08 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Knee Pain Chronic; Knee Osteoarthritis; Cartilage Damage; Cartilage Defects of the Knee; Cartilage or Osteochondral Defects in the Knee; Cartilage Lesion
Keywords: articular cartilage; cartilage lesion; focal cartilage defect; cartilage defect
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: randomized 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Investigational (Active Comparator): BioPoly Knee device
  Interventions: Device: BioPoly
- Control (Active Comparator): Surgical Standard of Care Group: either Microfracture or debridement procedure
  Interventions: Procedure: surgical standard of care (SSOC)

INTERVENTIONS:
Device: BioPoly — partial resurfacing knee replacement
  Arms: Investigational
Procedure: surgical standard of care (SSOC) — either microfracture or debridement
  Arms: Control

SUMMARY:
The goal of this randomized controlled clinical trial is to demonstrate the safety and effectiveness of the BioPoly® Partial Resurfacing Knee Implant for the treatment of cartilage defects of the distal femur in adult patients with knee pain and symptoms who are candidates for surgical intervention of the knee compared to outcomes for the control group.

The primary effectiveness endpoint is Month 24 composite clinical success (CCS) defined by:

* no secondary surgical intervention (SSI) and
* an improvement from baseline in the Knee injury and Osteoarthritis Outcome Score (KOOS) total score (scaled 0 to 100) of at least 10 points.

Researchers will compare the CCS for the investigational device group to a control group receiving the standard of care, either microfracture or debridement).

Subjects randomized to the investigational group will receive the BioPoly Knee device and those randomized to the control group will receive the current standard of care, either microfracture or debridement.

DETAILED DESCRIPTION:
The BioPoly® Partial Resurfacing Knee Implant is a surgical intervention when conservative therapies have been ineffective for focal cartilage lesions in the femoral condyles and is an early intervention prior to partial or total joint replacement. It is indicated for focal lesions with healthy surrounding and opposing cartilage. Specifically, the BioPoly® device is intended for the replacement of symptomatic abnormal or severely abnormal (ICRS Grade 2, 3 or 4) chondral or osteochondral focal lesions located in the femoral condyles or trochlear facets in patients between 30 and 65 years of age.

The RCT compares the primary endpoint, Composite Clinical Success criteria, for the investigational device, the BioPoly device, to that of the control group, which is the standard of care for these focal lesions either microfracture or debridement.

For those patients who meet eligibility criteria, randomization is 1:1. For the control group, there is a treatment algorithm to determine if microfracture or debridement that is based upon age of the subject, Kellgren-Lawrence score, and lesion size.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is between 30 and 65 years of age25.
2. KOOS quality of life score ≤ 60.
3. In the opinion of the Investigator, the patient has the understanding and willingness to comply with all study requirements including the Post-Operative rehabilitation and follow-up protocol.
4. Patient has cartilage lesion that has failed non-surgical conservative therapy (e,g, anti-inflammatory (NSAID), viscosupplementation, steroid injection, physical therapy, or activity modification) after at least 2 months of beginning the therapy or failed surgical conservative therapy (e.g. debridement/lavage, marrow stimulation, or alignment high tibial osteotomy) that was performed at least 12 months ago in the index knee and is a candidate for surgical intervention.
5. Patient has cartilage lesion located in the femoral condyle or trochlear facet.
6. Patient has lesion(s) classified as ICRS grade 2, 3 or 4.
7. Patient's lesion size may not exceed 3.1 cm2 and must be circumscribed by a 1.5 cm or 2.0 cm diameter circle, or 1.5 cm (M-L) by 2.4 cm (A-P) oval of normal or nearly normal (ICRS grade 0 or 1) cartilage, with an overall depth less than 4mm from the articulating surface.
8. Patient has subchondral bone quality that is non-osteoporotic and is sufficient to support the implant. The quality of bone will be assessed by the surgeon intraoperatively with a surgical instrument such as an awl.

Exclusion Criteria:

1. Patient has body mass index (BMI) ≥ 35.
2. Patient has autoimmune arthritis, as diagnosed by Investigator.
3. Patient has advanced degenerative osteoarthritis in index knee (Kellgren-Lawrence Grade 4 and/or diagnosed intraoperatively).
4. Contralateral knee is known to have symptomatic cartilage, meniscal, or ligamentous lesions, generalized osteoarthritis, or requires surgery.
5. Patient has gout, by Investigator diagnosis or patient-reported history within last 12 months.
6. Patient has a cartilage lesion that is being treated with a non-surgical conservative therapy (e,g, anti-inflammatory (NSAID), viscosupplementation, steroid injection, physical therapy, or activity modification) and it has been < 2 months since beginning treatment or the patient's cartilage lesion has failed surgical therapy (e.g. debridement/lavage, marrow stimulation, alignment (high tibial osteotomy)) in the index knee and it has been < 12 months since the surgical treatment.
7. Patient has a cartilage lesion that is being treated that has failed ACI, OATS or Allograft treatment.
8. Patient has malalignment of the index knee (>5 degrees weight bearing varus or valgus).
9. Patient has bipolar articular cartilage involvement (or kissing lesions) of the ipsilateral compartment (i.e. greater than ICRS Grade 2 on the opposing articular surface) in the index knee.
10. Patient has uncorrected ligamentous instability (good joint stability in the index joint with a Grade 1 Lachman or less, no pivot shift for ACL insufficiency and no posterior translation of more than grade 1; no deficits in flexion or extension of > 10 degrees compared to contralateral knee) in the index knee.
11. Patient has undergone a total meniscectomy of index knee.
12. Patient has undergone patellofemoral arthroplasty of the index knee
13. Patient currently reports or has a documented history of uncontrolled diabetes.
14. Patient currently has any condition, therapy, or medication known to impair bone healing.
15. Patient has had an active systemic infection or joint infection in index knee over the last 12 months.
16. Patient has an allergy to titanium alloy (Ti-6Al-4V), ultrahigh molecular weight polyethylene (UHMWPE), or hyaluronan/ hyaluronic acid (HA).
17. Patient is pregnant or is planning to become pregnant (for female patients only) at any point during the duration of the study.
18. Patient has legal involvement or any other issue that would hinder completion of the two-year follow-up period.
19. Patient is participating in other studies and/or receiving any other simultaneous therapy in index knee.
20. Patient has an uncorrected tear of the meniscus of the index knee. (Partial meniscectomy that retains >50% of the meniscus is allowed prior to or concurrently with the cartilage treatment procedure. Meniscus suture repair is allowed prior to or concurrently with the cartilage treatment procedure if >50% of the functional meniscus remains.).
21. Patient has an additional cartilage lesion(s) (ICRS Grade 3 or 4) in the index knee, located on the patella, trochlea, tibia, or non-weight bearing area of index condyle that requires treatment.
22. More than one implant is required to accommodate defect in the index knee.
23. Patient has inadequate bone stock (e.g., cysts, osteoporosis) underlying the lesion site as determined intra-operatively by the investigator

    1. As determined by the investigator through use of an awl or a similar instrument to determine if the bone quality is insufficient to support the BioPoly device.
    2. If the cause of inadequate bone stock is due to cysts or to the boney portion of an osteochondral lesion being excessive, then the investigator may opt to fix the implant with cement rather than exclude the patient for inadequate bone stock.
24. Patients with osteoporosis, osteopenia, Paget's disease, osteomalacia or any other metabolic bone disease; a. Osteoporosis is defined as Simple Calculated Osteoporosis Risk Estimation (SCORE) above 6 and DXA T-score < -2.5 or QCT T-score < 80mg/cubic cm. History of a fragility fracture requires that a DXA scan or QCT scan is completed

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in the Knee injury and Osteoarthritis Outcome Score (KOOS) to Assess Composite Clinical Success (CCS) effectiveness | 24 months
  An improvement from baseline in the Knee injury and Osteoarthritis Outcome Score (KOOS) total score (scaled 0 to 100) of at least 10 points. If this criteria is met, the subject will be considered as a success relative to the measure of the Clinical Composite Success for effectiveness.
Composite Clinical Success (CCS) Safety as Measured by No Secondary Surgical Intenvention | 24 months
  No secondary surgical intervention (SSI) by 24 months will be considered as a success for the subject relative to the Composite Clinical Success (CCS) for Safety.

SECONDARY OUTCOMES:
Effectiveness over 24 months as measured by the Knee injury and Osteoarthritis Outcome Score (KOOS) | 24 months
  KOOS individual component sub-scales (Pain, Symptoms, Activities of Daily Living, Sports/Recreation, Quality of Life) as measured by change from baseline at 6 weeks, 3, 6, 12, and 24 months. The minimum and maximum raw scores for each sub-scale is as follows: Pain = 0-36, Symptoms = 0-28, Activities of Daily Living = 0-38, Sports/Recreation = 20, Quality of Life = 0-16. The sub-scales will be reported on a normalized scale relative the maximum raw score for the particular sub-scale, thus, each sub-scale score will have a range of 0-100 with 100 being better. For instance, a subject's Quality of Life raw score of 12 would be normalized as 12/16 x 100 = 75 points. The reported number will be the difference between the normalized score at a particular timepoint minus the baseline normalized score.
Effectiveness pain reduction over 24 months | 24 months
  Variable Analog Scale (VAS) Pain score as measured by change from baseline at 6 weeks, 3, 6, 12, and 24 months. The VAS Pain score ranges from 0-100 where a lower number is a measure of less pain; so, lower VAS Pain scores are better.
Adverse Events Over 24 Months | 24 months
  * Serious device-related adverse events through 24 months
  * Device-related adverse events through 24 months
  * Serious adverse events through 24 months
  * Unanticipated adverse device effects (UADE) through 24 months
Radiograph review to Assess Implant Stability Over 24 Months | 24 months
  Implant stability over time is assessed by monitoring implant migration/subsidence, implant loosening, and radiolucencies around the implant at 24 months.
Survival Over 24 Months | 24 months
  A survival analysis will be performed to determine the number of treated and control subjects that did not have a secondary surgical intervention to remove the implant or to perform another procedure to treat the same cartilage lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Herb Schwartz, Ph.D., Study Director — BioPoly LLC
Locations (1):
- Dupont Hospital, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Sharing of any data will only be in the aggregate.